CLINICAL TRIAL: NCT01460017
Title: Comparison Between The Outcome of Deep Sclerectomy and Traditional Trabeculotomy and Trabeculectomy Surgeries in Congenital Glaucoma
Brief Title: Comparison Between Deep Sclerectomy and Traditional Trabeculotomy & Trabeculectomy in Congenital Glaucoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Dr. Ahmed Mousa, Lecturer, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-11-487
Record Dates: First submitted 2011-10-25; First posted 2011-10-26 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Congenital Glaucoma
MeSH Terms: conditions — Hydrophthalmos

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS arm (Active Comparator): Deep sclerectomy surgery will be conduct in this arm
  Interventions: Procedure: Deep Sclerectomy
- Trab arm (Active Comparator): combined Trabeculectomy and Trabeculotomy surgery will be conducted in this arm
  Interventions: Procedure: Combined Trab

INTERVENTIONS:
Procedure: Deep Sclerectomy — Non penetrating glaucoma surgery is a new procedure in adults that has less post operative complications with good results, it is to be applied in children.
  Other Names: Non penetrating DS
  Arms: DS arm
Procedure: Combined Trab — Combined trabeculectomy and trabeculotomy is a standard surgery for congenital glaucoma, however, it has its known complications.
  Other Names: Combined Trabeculectomy Trabeculotomy
  Arms: Trab arm

SUMMARY:
The investigators hypothesize that deep sclerectomy in congenital glaucoma is a safer procedure and may yield better results than trabeculotomy trabeculectomy approach.

DETAILED DESCRIPTION:
Non penetrating glaucoma surgery depends on filtration through trabeculo-descmeto window as well as supra-choroidal space less to sub-conjunctival rout. the nature of the operation keeps the globe intact without penetration that leads to less complications compared to penetrating trabeculectomy combined with trabeculotomy.

ELIGIBILITY:
Inclusion Criteria:

* Any case diagnosed as congenital glaucoma with enlarged corneal diameter more than 11 mm and intra-ocular pressure above 21 mmHg, including corneal edema or Habb's Stria with or without optic disc cupping.
* Any case diagnosed as primary or secondary congenital glaucoma to ocular or systemic abnormalities.
* Within the age of (0 - 12).

Exclusion Criteria:

* Cases of congenital glaucoma with previous intervention.
* Age above 12 Yrs.
* Cases with secondary glaucoma caused by surgical intervention, ocular co-morbidity, medications or trauma

Ages: 1 Day to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
reduction in IOP | 6 month
  decrease in the intraocular pressure to the normal limit (<22 - >6) mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Saleh A. Al-Obeidan, MD, Principal Investigator — King Saud University
Locations (1):
- King Abdul Aziz University Hospital, Riyadh, Riyadh Region, Saudi Arabia